CLINICAL TRIAL: NCT06587607
Title: Exploring Virtual Reality Mindfulness Training for Veterans With SCI and Chronic Pain
Brief Title: VR Mindfulness Training for Veterans With SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B4813-M; 1IK1RX004813 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury; Chronic Pain
Keywords: Spinal Cord Injuries; Chronic Pain; Virtual Reality; Mindfulness
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single non-randomized group will be used to gather evaluation data on needed modifications to enhance program fit to the SCI population needs to develop a tailored curriculum for SCI. Outcomes will involve pre-post evaluation of measures to determine if there are any direct or indirect impacts of the mindfulness program as a preliminary feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VA CALM (Experimental): This group will receive the VA CALM mindfulness programming.
  Interventions: Behavioral: VA Compassionate Awareness Learning Module (VA CALM) a mindfulness curriculum.

INTERVENTIONS:
Behavioral: VA Compassionate Awareness Learning Module (VA CALM) a mindfulness curriculum. — VA CALM is a 9 week mindfulness curriculum typically delivered at a once/week module pace in group settings during sessions that last approximately 60-90 minutes. Module topics include: Program Introduction, Why mindfulness, Perception, What Makes Something a Pleasant Experience?, Being Stuck, Getting Unstuck, Communication, Mindfulness in Daily Life, and Today is the First Dat of the Rest of Your Life.
  Other Names: VA CALM

SUMMARY:
This study involves delivering a mindfulness program that was developed for Veterans called VA Compassionate Awareness Learning Module (VA CALM) to Veterans with spinal cord injuries (SCI) to develop accommodations to make the VA CALM program more accessible for those with SCI. It will involve delivering the unmodified curriculum to a group of Veterans with SCI first to determine what areas need accommodations, working with a group of stakeholders to develop appropriate accommodations, and then delivering 1-2 modified modules via virtual reality to evaluate whether using virtual reality was feasible and acceptable for this program.

DETAILED DESCRIPTION:
The objectives of this study are to explore the feasibility and acceptability of a spinal cord injury (SCI) tailored, evidence-based mindfulness group known as VA Compassionate Awareness Learning Module (VA CALM) when delivered via virtual reality (VR) The project will first assess modification needs for SCI and then explore the feasibility and acceptability of delivering VA CALM-SCI over VR.

The long-term goals and significance of this study include studying the efficacy of VA CALM-SCI for the treatment of chronic pain and examining the comparative effectiveness between VR and video telehealth modalities to build evidence for the modified intervention. This work has the potential to improve care for Veterans with SCI who are at risk of being left out of innovative clinical advancements that improve quality of life and well-being, due to the complexity of their medical condition.

Aim 1: Conduct a formative evaluation of the VA CALM program to develop accommodations to improve program accessibility and acceptability for Veterans with SCI and chronic pain (VA CALM-SCI).

* Aim 1a: Deliver the VA CALM program to 10 Veterans with SCI over telehealth to conduct a formative evaluation of the VA CALM curriculum to tailor for SCI contextual needs.
* Aim 1b: Assemble a Steering Committee of SCI stakeholders (10 members) to develop appropriate strategies, accommodations, and recommended tools to support the delivery of VA CALM-SCI.

Aim 2: Explore the feasibility and acceptability of delivering VA CALM-SCI over a Virtual Reality platform for Veterans with SCI and chronic pain.

* Aim 2a: Assess potential VR applications and settings for delivery and testing of VA CALM-SCI.
* Aim 2b: Deliver 2 VA CALM-SCI modules over VR to Veterans with SCI to assess the feasibility and acceptability of using VR in this population to deliver mindfulness training.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Diagnosis of spinal cord injury with incomplete or complete tetraplegia based on AIS score OR incomplete or complete paraplegia based on AIS score.
* Endorses chronic pain lasting 3 months;
* age 18+ years
* Access to high-speed internet
* Endorse being (at least) minimally proficient on the computer (eg, able to check emails, read the news, etc.); be able, either independently or with caregiver support, to get online for virtual meetings and don/doff VR equipment
* Able to speak clearly and independently to participate in focus group interviews.

Exclusion Criteria:

-Individuals unable to consent for research or medical care are ineligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Mindfulness- Five Facet Mindfulness Questionnaire (FFMQ) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 1 Maximum Score: 5 Score Interpretation: Items are aggregated and averaged. Higher scores indicate greater mindfulness.
Pain- PROMIS-Pain Numeric Rating Scale (NRS) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 0 Maximum Score: 10 Score Interpretation: Single item measure, higher scores indicate greater pain intensity.
Mindfulness- Mindfulness Attention Awareness Scale (MAAS) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 1 Maximum Score: 6 Score Interpretation: Items are aggregated and averaged. Higher scores indicate greater mindfulness
Pain Interference- PROMIS-Pain Interference (PROMIS-PI, SF8a) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 8 Maximum Score: 40 Score Interpretation: Scores are converted into a T-score which rescales the score into a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate greater pain interference.
Pain Acceptance- Chronic Pain Acceptance Questionnaire-Revised (CPAQ-R) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 0 Maximum Score: 6 Score Interpretation: Generates scores for two domains: Activity Engagement and Pain Willingness. Scores for each item in a domain are aggregated. Higher scores indicate higher levels of acceptance.
Pain Catastrophizing- Pain Catastrophizing Scale (PCS) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 0 Maximum Score: 52 Score Interpretation: Generates a total score PCS-T and three subscale scores: Rumination, Magnification, and Helplessness. Total score above 30 indicates clinically relevant level of catastrophizing.

SECONDARY OUTCOMES:
Quality of Life- World Health Organization Quality of Life-Brief (WHOQOL-BREF) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 4 Maximum Score: 20 Score interpretation: Measure is comprised of 4 quality of life domains: physical health, psychological health, social relationships, and environment. Items for each domain are aggregated, averaged, then scaled for final scoring. Higher scores indicate higher quality of life.
Anxiety- Generalized Anxiety Disorder (GAD-7) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 0 Maximum Score: 21 Score Interpretation: Higher scores indicate more severe anxiety. 0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, 15-21: severe anxiety.
Depression- Patient Health Questionnaire-9 (PHQ-9) | Baseline to 2 weeks post completion (Approx 14 weeks).
  Minimum Score: 0 Maximum Score: 27 Score Interpretation: Item scores are aggregated. Higher scores indicate greater depression severity. 0: no depression, 1-4: minimal depression, 5-9: mild depression, 10-14: moderate depression, 15-19: moderately severe depression, 20-27: severe depression.
Virtual Reality Embodiment- One-Item Presence Scale | After completion of 2nd VR session (One time point at completion of study, approximately week 12).
  Minimum Score: 1 Maximum Score: 10 Score Interpretation: Single item. Higher score indicates greater virtual presence.
Virtual Reality Embodiment- Virtual Embodiment Questionnaire | After completion of 2nd VR session (One time point at completion of study, approximately week 12).
  Minimum Score:1 Maximum Score: 7 Scoring interpretation: Measures 3 domains: Acceptance (ownership), Control (agency), and Change (perceived change in the body scheme). Item scores are aggregated then averaged for each domain. Higher scores indicate greater embodiment.
Acceptability of Virtual Reality- System Usability Scale (SUS) | After completion of 2nd VR session (One time point at completion of study, approximately week 12).
  Minimum Score: 0 Maximum Score: 100 Score interpretation: Items aggregated. Higher scores indicate greater usability.
Acceptability of Virtual Reality- Standardized User Experience Percentile Rank Questionnaire (SUPRQ) | After completion of 2nd VR session (One time point at completion of study, approximately week 12).
  Raw component Minimum Score: 1 Raw component Maximum Score: 5
  Percentile Minimum Score: 0 Percentile Minimum Score: 100
  Score interpretation: Two scores are generated and evaluated: Raw component score (1-5) which is aggregated and then averaged and percentile score (0-100). Higher scores indicate better user experience for both scales.
Acceptability of Program- Acceptability of Intervention Measure (AIM) | After completion of 2nd VR session (One time point at completion of study, approximately week 12).
  Minimum Score: 1 Maximum Score: 5 Score interpretation: Items aggregated then averaged. Higher scores indicate greater acceptability.
Acceptability of Program- Intervention Appropriateness Measure (IAM) | After completion of 2nd VR session (One time point at completion of study, approximately week 12).
  Minimum Score: 1 Maximum Score: 5 Score interpretation: Items aggregated then averaged. Higher scores indicate greater appropriateness.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Touchett, PhD MSN BSN, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in articles to be published after de-identification (text, tables, figures, and appendices) as required by publishers, funding agencies, and or by law.
  Further, a Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 36 months following article publication.
Access Criteria: Data sharing will be permitted for the purposes of validation of results via replication of analyses with the limited, de-identified database. Individually identifiable information will be removed from any database shared to ensure protection of personal privacy. Further the data will be shared pursuant to a data use agreement which prohibits re-identification.